CLINICAL TRIAL: NCT04131361
Title: Ultrasound-guided Inferior Vena Cava Diameter Dependent Colloid Challenge Versus Routine Crystalloid Strategy Fluid Replacement in Transurethral Resection Prostate (TURP) Under Spinal Anesthesia; A Prospective Randomized Controlled Study.
Brief Title: Inferior Vena Cava Diameter Dependent Colloid Challenge Versus Routine Crystalloid Strategy Transurethral Resection Prostate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mohamed Abd Latif Ghanim, Associate Professor os anesthesia ICU & Pain medicine., Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: R.19.10.644
Record Dates: First submitted 2019-10-12; First posted 2019-10-18 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Volume Overload
MeSH Terms: conditions — Edema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Crystalloid -control group: (Active Comparator)
  Interventions: Other: Ultrasound-guided Inferior vena cava diameter dependent colloid challenge versus routine crystalloid strategy Fluid replacement
- Colloid- study group: (Experimental)
  Interventions: Other: Ultrasound-guided Inferior vena cava diameter dependent colloid challenge versus routine crystalloid strategy Fluid replacement

INTERVENTIONS:
Other: Ultrasound-guided Inferior vena cava diameter dependent colloid challenge versus routine crystalloid strategy Fluid replacement — The inferior vena cava largest and smallest diameters will be measured proximal to the opening of the hepatic veins in the longitudinal axis with the M-mode using a 8-2 MHz curved array ultrasound probe placed longitudinally in the subcostal region.

SUMMARY:
Background: Intravenous fluid replacement during transurethral resection of the prostate is still unclear. Ultrasonography of the inferior vena cava (IVC) has been recently used to assess the volume status and predict fluid responsiveness. In this double-blind, randomized controlled study, we will assess the IVC at baseline and at subsequent time points after spinal anesthesia, and according to IVC diameter will give the replacement challenge colloid. Potential problems during TURP are mostly due to either fluid overload or bleeding: Intraoperative TURP syndrome, Hemorrhage, Myocardial ischemia, Hypothermia, Prostatic capsular perforation, Bladder or urethral perforation. Postoperative TURP syndrome, myocardial ischemia/infarction, Postoperative cognitive impairment. Study Hypothesis: Strict colloid volume optimization using US-guided IVC diameter calculation aiming decrease the total IV fluid volume and accommodate the transurethral inevitable absorption of currently used irrigation crystalloid fluid (Nacl0.9%) that accidentally absorbed and change it from a circulatory overload to a complementary part of the replacement IV fluids preventing fluid overload and TURP syndrome. Aim of the work: To reduce Intraoperative and postoperative fluid overload during TURP surgery with hemodynamic stability relaying up on US-guided IVC diameter dependent Strict IV Colloid replacement volume optimization. Methods: A prospective randomized controlled trial on ASAI-III male patient aged 40-80 years old subjected to transurethral endoscopic resection of the prostate (TURP) surgery. Then patients will be divided into 2 groups according to the IV infusion fluid type as follow: Crystalloid -control group: (preload plus continuous IO Ringer acetate crystalloid 4/2/1 rule infusion) according to the usual 4/2/1 rule. Not guided by IVC diameter but IVC diameter will be calculated using the US and recorded at baseline just after spinal anesthesia and then every 30 minutes till the end of surgery. Loop Diuretic (Furosemide) will be given according to the maximum diameter of the IVC as follow; 10mg if IVC>2.5Cm. Colloid- study group: (preload plus colloid challenge only); Fluid challenge boluses of 250 mL (over 5 minutes using a pressurizer) 6% hydroxyethyl starch 130/0.4 in 0.9% sodium chloride (voluven®) if the IVC<1.7(higher limit of normal) will be given guided by IVC diameter at baseline just after spinal anesthesia and then every 30 minutes till the end of surgery.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria:

  * Patients subjected to transurethral resection of prostate TURP.
  * ASA I&II
  * Age 40-80years old. prostate size 45-100
  * Surgical procedure: laser and Bipolar TURP using saline 0,9% irrigation.
* Exclusion Criteria:

  * Height <150 cm.
  * Weight <60 kg.
  * Body mass index ≥45 kg/m2.
  * Contraindications to spinal anesthesia (increased intracranial pressure or local skin infection).
  * Uncontrolled; Diabetes mellitus, cardiovascular failure, cerebrovascular uncontrolled deficite, or other renal disease.
  * Hemoglobin <10 gm/dL.
  * International Normalized Ratio >1.4
  * Platelet count <100,000 /mm3.
  * Preoperative serum creatinine >1.5 mg/dL

Ages: 40 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 34 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
total iv fluids | just after end of surgery

SECONDARY OUTCOMES:
serum Na at end of surgery | just after end of surgery
serum K at end of surgery | just after end of surgery
ximum and minimum IVC diameter | serial during surgery
IVC-CI | serial during surgery
Incidence of bradycardia | serial during surgery
Incidence of hypo-tension | serial during surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesia Department, Al Mansurah, Dakahlia Governorate, Egypt